CLINICAL TRIAL: NCT04407013
Title: Enhanced Supportive Care for Advanced Cancer Patients: Evaluation of Standardized Care Pathway
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4-2020-0304
Record Dates: First submitted 2020-05-18; First posted 2020-05-29 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Experimental group with application of the standardized care pathways and symptom management education
  Interventions: Other: Enhanced supportive care based on standardized care pathway
- B (Other): Control group with usual care (symptom monitoring only)
  Interventions: Other: Control group with usual care

INTERVENTIONS:
Other: Enhanced supportive care based on standardized care pathway — Enhanced supportive care based on standard care pathway is consisted of 1) symptom management (symptom assessment and according management) and 2) coping enhancement (nurse-led counseling). The enhanced supportive care will be provided 5 times, according to the standardized care pathway.
  Arms: A
Other: Control group with usual care — Control group will receive usual care (symptom monitoring only)
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the efficacy of the standardized care pathway which provides enhanced supportive care for patients with advanced cancer.

A pilot study (single arm pre-post test) will be conducted to evaluate feasibility of applying standardized care pathway to provide enhanced supportive care. A Randomized Controlled Trial will be conducted by randomly allocating participants in a 1:1 ratio to intervention arm (receiving enhanced supportive care according to the standardized care pathway) or control arm (receiving usual care: symptom monitoring only). Participants in the intervention arm will receive enhanced supportive care consisted of symptom management and coping enhancement counseling for 5 times. Data from advanced cancer patients will be collected at baseline (before start of chemotherapy), during chemotherapy (intervention arm), at the visit for cycle 5 of chemotherapy, at 6 month, and at 12 month Data from caregivers will be collected at baseline, 3 month, and 6 month. Primary outcomes will be measured as advanced cancer patients' symptom, coping and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* adult (age >=19 years old),
* cancer patients and their family
* ECOG =<2

Exclusion Criteria:

* patients with cognitive or psychiatric issue

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Symptom measured by the ESAS (Edmonton Symptom Assessment Scale + 5 additional symptoms) | at the visit for cycle 5 (each cycle is from 2 weeks to 4 weeks depending on chemotherapy regimen) of chemotherapy (at average 3 month)
Coping measured by brief COPE | at the visit for cycle 5 of chemotherapy (at average 3 month)
Quality of life measured by the EORTC QLQ C-30 | at the visit for cycle 5 of chemotherapy (at average 3 month)

SECONDARY OUTCOMES:
Depression measured by the HADS (Hospital Anxiety and Depression Scale) : research participation | at the visit for cycle 5 of chemotherapy (at average 3 month)
Depression measured by the HADS (Hospital Anxiety and Depression Scale) : research participation | at 6 month
Depression measured by the HADS (Hospital Anxiety and Depression Scale) : caregiver | at the visit for cycle 5 of chemotherapy (at average 3 month)
Depression measured by the HADS (Hospital Anxiety and Depression Scale) : caregiver | at 6 month
Self-efficacy measured by the Cancer Behavior Inventory 3.0 | at the visit for cycle 5 of chemotherapy (at average 3 month)
Self-efficacy measured by the Cancer Behavior Inventory 3.0 | at 6 month
Survival | at 6 month
Survival | at 12 month
Symptom measured by the ESAS (Edmonton Symptom Assessment Scale+5 additional symptoms) | at 6 month
Coping measured by brief COPE | at 6 month
Quality of life measured by the EORTC QLQ C-30 | at 6 month
Symptom change measured by the ESAS (Edmonton Symptom Assessment Scale + 5 additional symptoms): from baseline to 3 month | At baseline, at the beginning of Cycle 2, Cycle 3, Cycle 4, Cycle 5 (each cycle is from 2 weeks to 4 weeks depending on chemotherapy regimen)(at average 3 month)
Depression change measured by the HADS (Hospital Anxiety and Depression Scale): from baseline to 3 month | At baseline, at the beginning of Cycle 2, Cycle 3, Cycle 4, Cycle 5 (each cycle is from 2 weeks to 4 weeks depending on chemotherapy regimen)(at average 3 month)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi YY, Hong B, Rha SY, Cho S, Lee HS, Lee J. The effect of nurse-led enhanced supportive care as an early primary palliative care approach for patients with advanced cancer: A randomized controlled trial. Int J Nurs Stud. 2025 Aug;168:105102. doi: 10.1016/j.ijnurstu.2025.105102. Epub 2025 May 1. PMID 40378811
- [Derived] Choi YY, Rha SY, Cho S, Lee HS, Hong B, Lee J. Enhanced supportive care for advanced cancer patients: study protocol for a randomized controlled trial. BMC Nurs. 2022 Dec 2;21(1):338. doi: 10.1186/s12912-022-01097-5. PMID 36461000